CLINICAL TRIAL: NCT05461781
Title: Distal Radial Access for Primary Percutaneous Coronary Intervention in STEMI Patients to Prevent Acute Radial Artery Occlusion
Brief Title: Distal Radial Access for Primary PCI in STEMI Patients to Prevent RAO
Acronym: RAPIDIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Luhe Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Beijing LH
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: radial artery occlusion; primary percutaneous coronary intervention; distal radial access; conventional transradial access
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, parallel randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- distal radial access (Experimental): Distal radial access for primary percutaneous coronary intervention in STEMI patients
  Interventions: Procedure: distal radial access
- conventional transradial access (Active Comparator): conventional transradial access for primary percutaneous coronary intervention in STEMI patients
  Interventions: Procedure: conventional transradial access

INTERVENTIONS:
Procedure: distal radial access — primary percutaneous coronary intervention via distal radial access
  Arms: distal radial access
Procedure: conventional transradial access — primary percutaneous coronary intervention via conventional transradial access
  Arms: conventional transradial access

SUMMARY:
Randomized-controlled trial to compare early radial artery occlusion via distal vs. conventional transradial access among ST segment elevation myocardial infarction patients for primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
Conventional transradial access (TRA) is recommended as the default approach for patients undergoing percutaneous coronary intervention (PCI) according to 2018 ESC guidelines. However, radial artery occlusion (RAO) remains the frequent complication, precluding the future use of the radial artery as an access point for repeat coronary recanalization or as a conduit for coronary artery bypass surgery. More than 50% of patients with ST segment elevation myocardial infarction (STEMI) present multiple vascular lesions, of which 50% require reprocessing non-culprit vessels. Therefore, the patency of the radial artery is crucial for STEMI patients. The distal radial access (DRA), located in the anatomical snuffbox or the dorsum of the hand, was introduced as a promising alternative. Three recent RCTs have shown significant reductions of RAO after DRA compared with TRA. Nevertheless, all of them excluded the patients presenting with STEMI. Therefore, we conduct a prospective, single-center, open-label randomized clinical trial to assess the superiority of preventing RAO at 24 h via DRA when compared TRA among STEMI patients for primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ST-segment elevation myocardial infarction for primary percuteous coronary intervention
* Palpable pulses on both access sites of the radial artery
* Informed consent

Exclusion Criteria:

* Thrombolysis before primary percutaneous coronary intervention
* Previous CABG or radio-cephalic fistula using radial artery
* Cardiogenic shock
* Severe arrhythmias
* Severe liver and kidney dysfunction
* Pregnancy
* Enrolment in another study within 1 month
* Inability to obtain written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
radial artery occlusion | at 24 hours after procedure
  The radial artery occlusion will be evaluated 24 hours after procedure by ultrasound.

SECONDARY OUTCOMES:
the rate of successful puncture | Immediately post-procedurally
  Successful puncture occurs when an introducer sheath can be properly placed through the punctured artery.
puncture time | Immediately post-procedurally
  The puncture time was defined as the time interval between local anesthesia induction and successful sheath insertion.
first medical contact to device (FMC2D) time | Immediately post-procedurally
  FMC2D time was defined as the time interval between the patient's initial contact with the first physician who made the diagnosis and the first angioplasty balloon inflation.
procedural time | Immediately post-procedurally
  Procedural time defined as the time interval between local anesthesia to sheath removal.
hemostasis time | at 24 hours after procedure
  Hemostasis time was defined as the time between sheath removal to complete hemostasis.
access-related complications | at 24 hours after procedure
  Access-related complications include AV fistula formation, pseudoaneurysm, and local haematoma.
hand function | 1 week after procedure
  Hand function was evaluated by QuickDASH questionnaire.
radial artery occlusion | 30days after procedure
  The radial artery occlusion will be evaluated 1 month after procedure by ultrasound.
radial aretry injury | Immediately post-procedurally
  Radial aretry injury including intimal tears, dissections, perforation and thrombosis was detected by optical coherence tomography.
major adverse cardiovascular events(MACE) | 30 days after procedure
  MACE was defined as all-cause death, any myocardial infarction, stroke and major bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Jincheng Guo, Study Chair — Beijing Luhe Hospital
Locations (1):
- Beijing Luhe hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Z, Wang Y, Song J, Wang S, Wang Y, Wu Y, Wang H, Liu Z, Yan R, Zhai G, Guo J. Distal radial access to prevent radial artery occlusion for STEMI patients (RAPID III): a randomized controlled trial. BMC Med. 2025 Mar 24;23(1):173. doi: 10.1186/s12916-025-04005-1. PMID 40128873